CLINICAL TRIAL: NCT02488486
Title: Postoperative Sedation After Cardiac Surgery: Pilot Study
Brief Title: Postoperative Sedation After Cardiac Surgery
Acronym: SEDCAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Intermediate analysis
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014/24; 2014-A00949-38 (Other: ANSM)
Record Dates: First submitted 2015-06-26; First posted 2015-07-02 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Surgery, Cardiac; Anesthesia
MeSH Terms: interventions — Propofol; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Automated postoperative sedation (Experimental): Postoperative sedation is provided automatically using a closed-loop system. Bispectral index is used as the input signal and an algorithm defines the appropriate concentrations of propofol and remifentanil. Adequate postoperative sedation is defined by a bispectral index between 40 and 60.
  Interventions: Device: Automated postoperative sedation; Drug: propofol; Drug: remifentanil

INTERVENTIONS:
Device: Automated postoperative sedation
  Other Names: algorithm is the property of Medsteer SAS
Drug: propofol
Drug: remifentanil

SUMMARY:
This pilot study evaluates the effectiveness of a closed-loop administration of propofol and remifentanil guided by the bispectral index for short-term sedation after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* consent for participation
* cardiac surgical procedure requiring postoperative sedation

Exclusion Criteria:

* pregnant women,
* neurological or muscular disorder
* high risk of revision surgery
* patients having required a redo operation if the postoperative period of sedation was less than 2 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2015-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Level of sedation | 6 hours
  Richmond Agitation-Sedation Scale measured until extubation

SECONDARY OUTCOMES:
Level of pain during sedation | 6 hours
  Behavioral Pain Scale measured until extubation
Changes in hemodynamics profile consecutive to a tracheal suctioning | 6 hours
Changes in Bispectral Index consecutive to a tracheal suctioning | 6 hours
Changes in Richmond Agitation-Sedation Scale consecutive to a tracheal suctioning | 6 hours
Changes in Behavioral Pain Scale consecutive to a tracheal suctioning | 6 hours
Changes in concentration of propofol consecutive to a tracheal suctioning | 6 hours
Changes in concentration of remifentanil consecutive to a tracheal suctioning | 6 hours
Delay before awakening | 6 hours
  Delay between the cessation of infusion of propofol and remifentanil and extubation.
Number of temporary or definitive interruptions of the automated administration of propofol and remifentanil | 6 hours
Calculation of indices of performance of the closed-loop system | 6 hours
Periods of electrical silence | 6 hours
  Number and duration of electroencephalographic periods of silence
Total amounts of propofol observed during sedation period | 6 hours
Total amounts of remifentanil observed during sedation period | 6 hours
Changes in calculated plasma concentrations of propofol including minimum concentrations and maximum values | 6 hours
Changes in calculated plasma concentrations of remifentanil including minimum concentrations and maximum values. | 6 hours
Hemodynamic status during the sedation period | 6 hours
  Evolution of hemodynamic parameters (composite)
Hemodynamic status during the sedation period | 6 hours
  Number of medical interventions
Level of consciousness after extubation | 6 hours
  Richmond Agitation-Sedation Scale assessed every hour for three hours after extubation
Pain after extubation | 6 hours
  Simple numerical scale from 0 (no pain) to 10 (worst possible) assessed every hour for three hours after extubation
Awareness standardized questionnaire | 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Ambroise Paré, Neuilly-sur-Seine, Hauts-de-Seine, France

REFERENCES:
- [Background] Le Guen M, Liu N, Bourgeois E, Chazot T, Sessler DI, Rouby JJ, Fischler M. Automated sedation outperforms manual administration of propofol and remifentanil in critically ill patients with deep sedation: a randomized phase II trial. Intensive Care Med. 2013 Mar;39(3):454-62. doi: 10.1007/s00134-012-2762-2. Epub 2012 Dec 6. PMID 23223772